CLINICAL TRIAL: NCT02559453
Title: A Randomized Trial Comparing the Outcomes for 2 Operations Versus ≥ 3 Operations in Infected Wounds Requiring Hospitalization
Brief Title: Outcomes for 2 Operations Versus ≥ 3 Operations in Infected Wounds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Christopher Attinger, M.D., Director of the Center for Wound Healing, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 121012014
Record Dates: First submitted 2015-09-23; First posted 2015-09-24 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Wound Infection
MeSH Terms: conditions — Wound Infection | interventions — Debridement

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 operations (Active Comparator): Subjects in this arm will receive a maximum of two surgical debridements of their wound.
  Interventions: Procedure: Debridement
- 3 or more operations (Active Comparator): Subjects in this arm will receive three or more surgical debridements of their wound.
  Interventions: Procedure: Debridement

INTERVENTIONS:
Procedure: Debridement — Removing dead tissue from infected wounds.

SUMMARY:
We have designed this study to determine whether performing two, compared with ≥3 operations has an effect on key clinical outcomes after discharge from the hospital of an infected wound that requires admission. Each arm of this study represents the two commonly practiced standard of care treatment plans for patients presenting with infected wounds. It is currently unknown which SoC option provides the best patient outcome.

DETAILED DESCRIPTION:
There is a lack of consensus about whether or not a patient with an infected wound requires more than 2 surgical procedures. For patients admitted for an infected wound this study will investigate whether 2, compared with ≥3, operative interventions results in better outcomes. All patients admitted for an infected wound will be assessed for eligibility in the study. If eligible, subjects will be randomized into Cohort A (2 operative visits) or Cohort B (≥3 operative visits). Subjects will then be followed during the hospitalization as well as 180 days post discharge.

A total of 250 subjects will be enrolled into this study. Two operations (n=125) will be compared with ≥3 operations (n=125) during the hospitalization. We will compare the following factors between the two treatment groups: length of hospital stay; readmission post-discharge; quality of life; proportion of wounds closed or covered with a graft; culture results; host factors; environmental factors post-hospital discharge; and, financial charges related to admission and readmission. We expect full enrollment to take 3 years in duration.

Debridement of the wound will be performed in the customary manner per SOC in the operating room. Prior to the start of the study, the surgeons performing the operations will be required to view a video that demonstrates the standardized debridement technique that will be utilized. The following is the standardized technique depicted in the video:

All wound surfaces will be painted with dye prior to debridement. Debridement involves the use of a scalpel, scissors, curette, rongeur, or hydro-surgery. A 2-3 millimeter skin edge around the perimeter of the wound will also be resected. All infected/nonviable tissue will be removed and all tissues with dye will be surgically removed. This includes decompression of any purulent material and excision of any indurated tissue (until tissue pliability is established). Nonviable tissue includes necrotic and fibrous tissue. Debridement will be performed until the there is bleeding on the wound base and perimeter.

ELIGIBILITY:
Inclusion Criteria:

* Infected wound requiring hospital admission
* Infected wound requiring an operative intervention
* Wound can be located anywhere on the body
* Patient able and willing to comply with all study requirements

Exclusion Criteria:

* Planned free tissue flap for soft tissue reconstruction
* Wound located over exposed joint implant
* Wound located over exposed hardware
* Disease or treatment causing substantial immunosuppression
* History of collagen vascular disease
* Transplant recipient
* Venous stasis ulcer
* Radiation-induced ulcer
* Contraindication for use of negative pressure wound therapy with instillation of normal saline
* Unable or unwilling to comply with study requirements

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2015-09; Primary Completion 2020-03 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Number of post-hospital discharge complications between subjects who received 2 versus 3 or more debridement operations prior to closure. | 180 Days

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Attinger, MD, Principal Investigator — MedStar Georgetown University Hospital

IPD SHARING:
Plan to Share IPD: No
Data was not collected for use in future research and will not be shared.